CLINICAL TRIAL: NCT04943029
Title: Induction Therapy With Chemoimmunotherapy Followed by Surgery for Unresectable Stage III Non-small Cell Lung Cancer: a Single-center, Single-arm, Prospective Clinical Study
Brief Title: Neoadjuvant Immunotherapy and Chemotherapy Followed by Surgery in Unresectable Stage Ⅲ NSCLC
Acronym: NEOSUN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEOSUN
Record Dates: First submitted 2021-06-18; First posted 2021-06-29 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-06

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Unresectable; Stage Ⅲ NSCLC; Neoadjuvant; chemoimmunotherapy; camerlizumab; PD-1; sugery
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — camrelizumab; spartalizumab; Pemetrexed; Carboplatin; Antineoplastic Agents; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1+Chemo+surgery+PD-1 (Experimental): Participants will receive neoadjuvant Carrelizumab plus double platinum based chemotherapy for 3 cycles, followed by surgical resection and adjuvant Carrelizumab for 16 cycles.
  Interventions: Drug: Carrelizumab; Drug: Pemetrexed (Nonsquamous NSCLC) or Nab-paclitaxel(Squamous NSCLC); Drug: Carboplatin; Procedure: Surgery

INTERVENTIONS:
Drug: Carrelizumab — Camrelizumab: 200mg, IV, day 1 of each 21-day cycle, neoadjuvant therapy : 3 cycles; Adjuvant therapy: 16cycles.
  Other Names: PD-1 antibody
Drug: Pemetrexed (Nonsquamous NSCLC) or Nab-paclitaxel(Squamous NSCLC) — Nab-paclitaxel: 260mg/m^2, IV, day 1 of each 21-day cycle, 3 cycles; Pemetrexed: 500 mg/m^2, IV, day 1 of each 21-day cycle, 3 cycles.
Drug: Carboplatin — Carboplatin was given dosed to an area under the serum concentration-time curve (AUC) of 5 i.v. on day 1 of each 21-day cycle for 3 cycles.
  Other Names: chemotherapeutic drug
Procedure: Surgery — Surgery must be done within the 4th-6th week from day 1 cycle 3 of neoadjuvant treatment (4-6 weeks after day 1 of cycle 3)

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Camrelizumab in combination with platinum doublet neoadjuvant chemotherapy before surgery [neoadjuvant phase], followed by Camrelizumab alone after surgery [adjuvant phase] in participants with unresectable stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
Concurrent chemoradiotherapy is the recommended therapeutic approach for patients with unresectable stage III non-small cell lung cancer(NSCLC), although surgery offers the chance of cure. With combined radiation and chemotherapy, the prognosis of unresectable stage III NSCLC remains poor. Immunotherapy combined with chemotherapy has been shown to be efficacious as treatment for advanced non-squamous non-small-cell lung cancer (NSCLC) without targetable genetic aberrations. Camrelizumab, a humanised monoclonal antibody against PD-1, has shown its efficacy in the treatment of advanced NSCLC. This study is to studying neoadjuvant camrelizumab plus double platinum based chemotherapy followed by surgery to see how well it works in treating patients with unresectable stage III NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided.
* Age 18-70 when signing the consent form, both male and female;
* The ECOG score is 0 or 1;
* Unresectable stage III non-small cell lung cancer confirmed by histopathology or cytology（III A-bulky N2, III B，IIIC）;
* Adequate hematological function, liver function and renal function;
* Female participants should not be pregnant or breast-feeding.

Exclusion Criteria:

* EGFR mutation or ALK mutation was positive;
* Previously received systemic anti-tumor therapy for non-small cell lung cancer;
* Subjects who have received chest radiotherapy in the past;
* Known human immunodeficiency virus (HIV) infection;
* Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease);
* Pregnancy or breast-feeding women;
* Ingredients mixed with small cell lung cancer patients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-20 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Major pathological response (MPR) rate | 1 year
  MPR rate is defined as the percentage of participants having ≤10% viable tumor cells in the resected primary tumor and all resected lymph nodes following completion of neoadjuvant therapy.

SECONDARY OUTCOMES:
Resectability rate | 1 year
  Resectability rate is defined as the percentage of patients who were able to undergo surgery after neoadjuvant therapy.
Percentage of incidence of adverse Events | approximately 16.5 months overall
  The incidences and types of adverse events that occur during neoadjuvant therapy and perioperative period (within postoperative 30 days and 90 days) will be evaluated according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
PFS | 2 year
  Progression free survival
OS | 2 year
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Yongde Liao, PhD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Wuhan Union Hospital, Wuhan, China

IPD SHARING:
Plan to Share IPD: No